CLINICAL TRIAL: NCT04497714
Title: Identifying Ultrasonic Diagnostic Characteristics of Cervical Lymphadenopathy: A Retrospective, Multicenter Study
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 研2020-539
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Lymph Node Disease; Ultrasound Therapy; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cervical lymph nodes tuberculosis: The patients with Cervical lymph nodes tuberculosis
  Interventions: Diagnostic Test: Ultrasonic image collection
- Cervical lymphoma: The patients with
  Interventions: Diagnostic Test: Ultrasonic image collection
- Cervical lymph node metastasis: The patients with
  Interventions: Diagnostic Test: Ultrasonic image collection
- Cervical Reactive hyperplasia: The patients with
  Interventions: Diagnostic Test: Ultrasonic image collection

INTERVENTIONS:
Diagnostic Test: Ultrasonic image collection — Ultrasonic image collection,consist of three static images and one dynamic image

SUMMARY:
The observed indexes of the four cervical lymph node diseases were identified by informatics methods, and the differences in the diagnosis of the four diseases were evaluated, so as to improve the clinical diagnosis rate and provide a research basis for the ultrasonic evaluation of the surgical indications of cervical lymph node diseases in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one of these four diseases

Exclusion Criteria:

* 1. Patients with severe heart and brain diseases and poor coagulation function. 2. Undiagnosed patients are not included in the statistical analysis. 3. Image distortion of CEUS acquisition cannot be analyzed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with one of these four diseases
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Cervical lymph nodes tuberculosis | through study completion, an average of 1 year
  It was identified as cervical lymph node tuberculosis by imaging observation
Cervical lymphoma | through study completion, an average of 1 year
  It was identified as cervical lymphoma by imaging observation
Cervical lymph node metastasis | through study completion, an average of 1 year
  It was identified as Cervical lymph node metastasis by imaging observation
Cervical Reactive hyperplasia | through study completion, an average of 1 year
  It was identified as Cervical Reactive hyperplasia by imaging observation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ultrasound, Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data(IPD) can be shared after the main unit publish articles
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: by request
Access Criteria: by request